CLINICAL TRIAL: NCT06107582
Title: Clinical Characteristics, Prognosis and Prognostic Model of Pediatric Immune Thrombocytopenia: a Prospective, Multicenter, Observational Cohort Study
Brief Title: Longitudinal Cohort of Pediatric Primary Immune Thrombocytopenia (ITP)
Status: Recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Beijing Children's Hospital (Other); Tianjin People's Hospital (Other); Henan Cancer Hospital (Other Government); Tianjin Medical University Second Hospital (Other); The First Affiliated Hospital of Xiamen University (Other); The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: IIT2023044
Record Dates: First submitted 2023-08-26; First posted 2023-10-30 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-12

CONDITIONS: Primary Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Primary Immune Thrombocytopenia: Immune thrombocytopenia (ITP) : defined according to the international working group criteria
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — The study will collect basic information, diagnostic and treatment information from medical records and use questionnaire to measure the exposure of patients, and prospectively follow-up to collect the prognosis information.

SUMMARY:
Immune thrombocytopenic purpura (ITP) is a kind of rare childhood disease that involve autoimmune destruction of platelets.The current Pediatric ITP cohorts are mostly based on single-center or multi-center cases, or cohorts with limited sample size in China. There is a lack of comprehensive and large-scale prospective cohort studies in pediatric ITP. The purpose of this study is to analyze the clinical characteristics of Pediatric ITP, the treatment methods, prognosis and prognostic model of these patients in China.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an organ-specific autoimmune disease, which is characterized by decreased platelet count and skin and mucosal bleeding. ITP is a kind of disease with increased platelet destruction and impaired platelet production caused by autoimmunity. Conventional treatment of adult ITP includes first-line glucocorticoid and immunoglobulin therapy, second line TPO and TPO receptor agonist, splenectomy and other immunosuppressive treatments (such as rituximab, vincristine, azathioprine, etc.). ITP is one of the most common hemorrhagic diseases. At present, the treatment response of ITP is not good, and a considerable number of patients need drug maintenance treatment, which seriously affects the quality of life of patients and increases the economic burden of patients. Longitudinal Cohort allows to describe the long-term clinical characteristics of pediatric ITP patients, to study the benefit-risk balance of treatments, including the growing development of targeted therapies and to analyze the prognostic factors and attempts to establish prognostic models.

The study will include pediatric patients diagnosed with primary immune thrombocytopenia in the investigating hospitals, and collect basic information, diagnostic and treatment information from medical records. The study will use questionnaire to measure the exposure of patients, and prospectively follow-up to collect the prognosis information.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-17 years old (including both ends), male and female;
* Diagnosis of ITP.

Exclusion Criteria:

* Secondary thrombocytopenia caused by various reasons, such as connective tissue disorders, bone marrow hematopoietic failure disease, myelodysplastic syndrome, malignancy, drugs, inherited thrombocytopenia, common variable immune deficiency, lymphoma, etc.;
* The expected follow-up period is less than 3 months.

Ages: 6 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Pediatric patients who were diagnosed with ITP in the investigating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 3 years
  Overall response rate defined as proportion of subjects with a platelet count ≥ 30 × 10^9/L and at least 2-fold from baseline without bleeding
Time to onset response | 3 years
  Time to onset response defined as the time needed for subjects to have a platelet count ≥ 30 × 10^9/L and at least 2-fold from baseline without bleeding
Duration of response | 3 years
  Duration of response defined as the longest duration for which the subject sustained a platelet count ≥ 30 × 10^9/L and at least 2-fold from baseline without bleeding
Sustained response rate | 3 years
  Sustained response rate defined as proportion of subjects who keep a platelet count ≥ 30 × 10^9/L and at least 2-fold from baseline without bleeding at 6, 12, 24, 36 months after initial administration of certain treatment in absence of rescue therapy
Emergency treatment | 3 years
  Percentage of subjects who received emergency treatment after initial administration of certain treatment
Number of subjects with clinically significant bleeding as assessed using the bleeding scale for pediatric patients with ITP after initial administration of certain treatment | 3 years
  Changes of the subjects' numbers in bleeding score after administration of certain treatment according to the reported bleeding scale for pediatric patients with ITP. The bleeding scale for pediatric patients with ITP is a measure of bleeding severity with the following grades: Grade 1 (minor) Minor bleeding, few petechiae (≤100 total) and/or ≤5 small bruises (≤3 cm in diameter), no mucosal bleeding；Grade 2 (mild) Mild bleeding, many petechiae (>100 total) and/or >5 large bruises (>3 cm in diameter), no mucosal bleeding；Grade 3 (moderate) Moderate bleeding, overt mucosal bleeding, troublesome lifestyle；Grade 4 (severe) Severe bleeding, mucosal bleeding leading to decrease in Hb>2 g/dL or suspected internal hemorrhage；
Number of subjects with clinically significant bleeding as assessed using the world health organization (WHO) bleeding scale after initial administration of certain treatment | 3 years
  Changes of the subjects' numbers in WHO bleeding score after administration of certain treatment according to the reported World Health Organization's Bleeding Scale. The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
Recurrence-free survival rate | 3 years
  Time from the start of treatment to the occurrence of a relapse or death event

SECONDARY OUTCOMES:
Incidence | 3 years
  The incidence of pediatric primary immune thrombocytopenia in China will be described
Distribution | 3 years
  The population characteristics of pediatric primary immune thrombocytopenia in China will be described
Prognosis related factors selected from transcriptome data | 3 years
  The prognosis related factors will be selected from transcriptome data and be used to establish prognosis prediction model
Prognosis related factors selected from proteomics data | 3 years
  The prognosis related factors will be selected from proteomics data and be used to establish prognosis prediction model
Prognosis related factors selected from metabolomics data | 3 years
  The prognosis related factors will be selected from metabolomics data and be used to establish prognosis prediction model
Prognosis related factors selected from microbiome data | 3 years
  The prognosis related factors will be selected from proteomics data and be used to establish prognosis prediction model
Incidence, severity, and relationship of treatment emergent adverse events after treatment | 3 years
  Incidence, severity, and relationship of treatment emergent adverse events after treatment will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital
Locations (1):
- Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, China